CLINICAL TRIAL: NCT06021418
Title: A Single Center, Randomized, Subject and Evaluator Blinded, Split-face, Pivotal Clinical Trial to Evaluate the Efficacy and Safety of DKB-119 in Crow's Feet
Brief Title: Efficacy and Safety of DKB-119 in Patients in Crow's Feet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DKB-119-MD-2
Record Dates: First submitted 2023-04-19; First posted 2023-09-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-04

CONDITIONS: Crow's Feet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: 1. Blind: Participant, Outcomes Assessor
  2. Un-blind: Investigator(Care Provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DKB-119 (Experimental): Injecting to one side crow's feet
  Interventions: Device: DKB-119
- Control (Active Comparator): Injecting to one side crow's feet
  Interventions: Device: DKB-119

INTERVENTIONS:
Device: DKB-119 — Experimental and Acitve Comparator are applied 4 times to each of crow's feet on both sides of the subject.

SUMMARY:
To prove the non-inferiority of DKB-119 by evaluating the injecting efficacy and safety DKB-119 and control for patients in crow's feet

DETAILED DESCRIPTION:
A single center, randomized, subject and evaluator blinded, split-face, pivotal clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Those who are over 19 under 70 ages.
* Those who score 2 or more in the LCL severity evaluation.
* Those who have visually symmetrical crow's feet on both sides.
* Etc.

Exclusion Criteria:

* Pregnancy and lactating women.
* Etc.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-09-08 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Crow's feet | 18 weeks
  Difference in improvement rate (percentage)

SECONDARY OUTCOMES:
Crow's feet | 8, 10 weeks
  Difference in improvement rate (percentage)
LCL(Lateral Canthal Line) Severity | 8, 10, 18 weeks
  Difference in improvement rate (percentage)
GAIS(Global Aesthetic Improvement Scale) | 8, 10, 18 weeks
  GAIS 5 point scale (minimum -1 to maximum 3 points, The higher the score, the better the value)

CONTACTS AND LOCATIONS:
Locations (1):
- Chungang-University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No